CLINICAL TRIAL: NCT02584790
Title: Using Narrow-band Imaging (NBI) Technique to Detect Post-radiotherapy Mucosal Residual Nasopharyngeal Carcinoma (NPC)
Brief Title: NBI to Detect Post-RT Mucosal Residual NPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Dr. Wong Kai Chuen, Doctor, Pamela Youde Nethersole Eastern Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NBI1782015
Record Dates: First submitted 2015-08-17; First posted 2015-10-23 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Narrow band imaging
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Laryngoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post radiotherapy 8 weeks NPC patient (Other): All post-radiotherapy 8 weeks NPC patient will routinely undergo laryngoscope examination (WL system) and NP biopsy will be taken at the same time to determine if there is any residual NPC. In this study, laryngoscope with NBI system will be used. NBI system will be turn on during the post radiotherapy 8 week laryngoscope examination in additional to routine WL system
  Interventions: Device: Laryngoscope with NBI system

INTERVENTIONS:
Device: Laryngoscope with NBI system — All post-radiotherapy 8 weeks NPC patient will routinely undergo laryngoscope examination (WL system) and NP biopsy will be taken at the same time to determine if there is any residual NPC. In this study, laryngoscope with NBI system will be used. NBI system will be turn on during the post radiotherapy 8 week laryngoscope examination in additional to routine WL system

SUMMARY:
NBI has been proven to be a useful tool to detect early NPC, but they were few studies concerning the detection of post-radiotherapy mucosal residual NPC using NBI system

DETAILED DESCRIPTION:
Background

NPC has a uniquely high prevalence in Southern China. According to the Hong Kong Cancer Registry in 2012, NPC was the sixth commonest cancer in men and thirteenth in women. It accounted for 2.9% of all new cancer cases. In 2012, there were 819 new cases of NPC.

NPC is highly radiosensitive. Radiotherapy and chemotherapy are the mainstay of treatment. Despite the chemo-irradiation, disease control failure still occurred in NPC patients presenting as persistent tumor. Early detection of those post-radiotherapy residual NPC is essential for early arrangement of salvage therapy. Detection methods include imaging, plasma Epstein-Barr virus DNA, endoscopy examinations and nasopharynx biopsy.

NBI system has been well proven as a tool to detect early digestive tract cancer and head and neck cancer. However, there were only few studies targeting the detection of post-radiotherapy mucosal residual of NPC using NBI system

Objective

1. To identify the vessel pattern of those confirmed NPC case using NBI system
2. To identify the endoscopy features of post-radiotherapy mucosal residual nasopharyngeal carcinoma using NBI system
3. To establish the positive predicted value, negative predicted value, sensitivity and specificity of using NBI system for detecting mucosal residual NPC

Method:

1. All newly biopsy confirmed NPC patient will be assessed, their nasopharynx endoscopic image will be captured using both WL + NBI system
2. At post-radiotherapy 8th weeks, endoscopic examination will be arranged for patient using both WL + NBI system, biopsy will also be taken to detect mucosal residual NPC

ELIGIBILITY:
Inclusion Criteria:

* all new NPC patient

Exclusion Criteria:

* History of radiotherapy to head and neck region
* Poor premorbid status/ non-communicable patients
* <18 years old
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wong Kai Chuen, MBChB, MRCS, Principal Investigator — Pamela Youde Nethersole Eastern Hospital
Locations (1):
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post Radiotherapy 8 Weeks NPC Patient
Started | 55
Completed | 40
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Post Radiotherapy 8 Weeks NPC Patient
Number analyzed (Participants) | 55
Age, Customized [Count of Participants; unit: Participants]
  < 18 years old | 0
  >= 18 years old | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 55
NPC patients [Count of Participants; unit: Participants] | 40

OUTCOME MEASURES:

1. Primary Outcome: Positive Nasopharynx Biopsy Results Detected by NBI System in Those Post-radiotherapy 8th Week NPC Patient
Description: 4 grading of NBI vessel patterns can be identified in those post-radiotherapy 8 weeks NPC patients.
  Grade A: normal vessel size and length, regular pattern Grade B: normal vessel size, short, regular spiderweb like pattern Grade C: irregular vessel size and length, distorted and irregular pattern Grade D: thickened vessel size, elongated, distorted, and earthworm pattern
Time Frame: Post-radiotherapy 8th week
Measure: Number; unit: participants
Arm/Group | Post Radiotherapy 8 Weeks NPC Patient
Number analyzed (Participants) | 40
participants
  Grade A, no residual NPC | 14
  Grade A, positive residual NPC | 1
  Grade B, no residual NPC | 20
  Grade B, positive residual NPC | 1
  Grade C, no residual NPC | 1
  Grade C, positive residual NPC | 1
  Grade D, no residual NPC | 1
  Grade D, positive residual NPC | 1

2. Secondary Outcome: Assocication of Residual NPC With NBI Non Suspicious Pattern Group and NBI Suspicious Pattern Group
Description: Non suspicious pattern = grade A + grade B Suspicious pattern = grade C + D
  The sensitivity, specificity, positive predicted valve and negative predicted valve of detecting mucosal residual NPC using NBI suspicious/ non suspicous pattern can be thus calculated.
Time Frame: Post-radiotherapy eight weeks
Population: NBI non suspicious pattern = 36 NBI suspcious pattern = 4 Total = 40
Measure: Count of Participants; unit: Participants
Arm/Group | Post Radiotherapy 8 Weeks NPC Patient
Number analyzed (Participants) | 40
Participants
  NBI non suspicious pattern: number analyzed (Participants) | 36
  NBI non suspicious pattern: without residual disease | 34
  NBI non suspicious pattern: with residual disease | 2
  NBI suspicious pattern: number analyzed (Participants) | 4
  NBI suspicious pattern: without residual disease | 2
  NBI suspicious pattern: with residual disease | 2
Statistical Analysis 1: Comparison: Post Radiotherapy 8 Weeks NPC Patient; 2x2 table of: Row: 1. NBI suspicious pattern 2. NBI non-suspicious pattern Category: 1. with residual disease 2. without residual disease; Test type: Other; p = 0.004, Chi-squared

3. Secondary Outcome: The Sensitivity, Specificity, Positive Predicted Valve and Negative Predicted Valve of Detecting Mucosal Residual NPC Using NBI Suspicious/ Non Suspicous Pattern
Description: as for outcome 2
Time Frame: Post-radiotherapy eight weeks
Population: NBI non suspicious pattern = 36 NBI suspcious pattern = 4 Total = 40
Measure: Number; unit: Percentage of participants
Arm/Group | Post Radiotherapy 8 Weeks NPC Patient
Number analyzed (Participants) | 40
Percentage of participants
  Sensitivity | 50
  Positive Predicted Valve | 50
  Specificity | 94
  Negative Predicted Valve | 94

ADVERSE EVENTS:
Time Frame: 1 year 2 months
Arm/Group | Post Radiotherapy 8 Weeks NPC Patient
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
Small sample size Observation bias Musosal trauma during endoscopy examination hinder vessel identification

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-11-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT02584790/Prot_000.pdf
  • Informed Consent Form (2015-11-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT02584790/ICF_001.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT02584790/SAP_002.pdf